CLINICAL TRIAL: NCT00357383
Title: Study of the Ocular Safety After Repeated Instillations of T1225 1% or 1.5% Eye Drops in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LT1225-PI3-07/02(F)
Record Dates: First submitted 2006-07-25; First posted 2006-07-27 (Estimated); Last update posted 2006-07-27 (Estimated); Status verified 2006-07

CONDITIONS: Eye Infections, Bacterial
MeSH Terms: conditions — Eye Infections, Bacterial | interventions — Azithromycin

INTERVENTIONS:
Drug: Azithromycin (T1225)

SUMMARY:
To evaluate the ocular tolerance of T1225 1% and 1.5% eye drops versus vehicle after one instillation twice-daily (morning and evening), in one eye, during 3 days (from Day 0 to Day 2).

To assess azithromycin tear, conjunctiva and plasmatic concentrations, after a 3-day treatment period

DETAILED DESCRIPTION:
The aim of the present study was to compare ocular tolerance and safety after repeated instillations of T1225 1% and 1.5% eye drops and vehicle and to assess the residual azithromycin concentrations in tear, ocular conjunctiva and plasma samples, approximately 12 hours after the last Investigational Medicinal Product instillation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged from 18 to 45 years old;
* Written informed consent;
* Healthy volunteers without any subjective ocular symptom;
* Normal ocular examination in both eyes (corrected visual acuity >= 6/10, normal slit lamp examination, tear prism height > 0.1mm, tear break-up time (BUT) >= 10 seconds, lissamine green test score < 4);
* Registered, or agreed to be registered, in the national register of healthy volunteers

Exclusion Criteria:

* Ocular trauma, infection or inflammation within the last 3 months;
* number of corneal stained punctuations Ocular trauma, infection or inflammation within the last 3 months;
* number of corneal stained punctuations >= 5;
* blepharitis, conjunctivitis, uveitis;
* contact lenses;
* topical ocular treatment within the last month;
* ocular laser within the last 3 months;
* ocular surgery, including LASIK and PRK, within the last 12 months;
* systemic macrolide within the last month;
* medication during the study (except: paracetamol and contraceptives).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2002-10; Study Completion 2002-10

PRIMARY OUTCOMES:
Ocular pharmacokinetic in tears

SECONDARY OUTCOMES:
Tolerance

CONTACTS AND LOCATIONS:
Overall Officials: Didier CHASSARD, Dr, Principal Investigator — ASTER, Paris, France